CLINICAL TRIAL: NCT02702804
Title: High Intensity Interval Training for People With Mild Multiple Sclerosis: A Feasibility Study
Acronym: HIIT-MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Sheffield Hallam University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STH18899
Record Dates: First submitted 2016-02-18; First posted 2016-03-09 (Estimated); Last update posted 2019-11-14 (Actual); Status verified 2018-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- High Intensity Interval Training (Experimental): Participants will attend two sessions per week for the 6 week intervention. Each session will consist of 6-10 sets of 60 second high intensity intervals interspersed with 60 seconds recovery. The workload during each interval will be set at 80-90% of peak power achieved during the VO2peak test. This is predicted to elicit 85-95% heart rate reserve in the participants. After each interval the participant's heart rate and rate of perceived exertion (RPE) will be collected. After each session a researcher will complete an Adverse Event form to record if an event occurred or not. Additionally the participant will complete a physical activity enjoyment (Perceived activity enjoyment scale) after one session per week.
  Interventions: Other: High Intensity Interval Training

INTERVENTIONS:
Other: High Intensity Interval Training — High Intensity Interval Training

SUMMARY:
Exercise has been shown to improve quality of life in people with multiple sclerosis but most exercise programmes are carried out at low to moderate intensities. The next stage in the management of the condition is to establish if people with mild Multiple Sclerosis can exercise, safely and effectively at a higher intensity. High intensity interval training (HIIT) involves repeated bursts of hard exercise interspersed with periods of rest. High intensity interval trainingcould be a time efficient and safe option for people with Multiple Sclerosis. Potential improvements are; cardiovascular fitness, resistance to fatigue, balance, quality of life and attitude to physical exercise.

Participants will attend two sessions per week for 6 weeks. Each session will involve 6-10 sets of 60 seconds of high intensity cycling followed by 60 seconds rest. Potential participants must have a clinical diagnosis of Mulitple Sclerosis for more than 3 months, an EDSS score of less than 2.5, aged 18-65, and had no more than one relapse in the last 2 years.

From this study the investigators hope to discover if High Intensity Interval Training is a safe and enjoyable form of physical activity for people with mild Multiple Sclerosis. This will then hopefully lead to further large research trials.

DETAILED DESCRIPTION:
Multiple Sclerosis is an autoimmune disease that is typically progressive and involves damage to the nerve cells in the central nervous system. Living with multiple sclerosis can be a difficult experience both physically and psychologically. Some of the most common symptoms for people with MS include excessive fatigue, limb weakness, motor abnormalities and sexual dysfunction with symptoms dependant on the central nervous system pathology. Multiple Sclerosis is the most common cause of disability in young to middle aged adults in the developing world. The relatively high incidence rates and longitudinal nature of the condition has a large economic impact on the health care system, people with Multiple Sclerosis and their families. Treatments are now able to better manage the condition but there is still no cure and the fundamental cause is still unknown, so symptom management and maintenance of function is crucial. Exercise and rehabilitation are increasingly being looked at to allow patients to better manage their condition and assist people with multiple sclerosis to self-manage their care.

For many years people with multiple sclerosis have limited their activity levels to in order to not exasperate their symptoms. Since then research has shown that supervised exercise (aerobic and strength) training can be beneficial for people with mild to moderate multiple sclerosis. Current evidence now suggests that exercise may actually go even further than improving function and better managing symptoms in multiple sclerosis, but may actually have a disease modifying effect, suggesting that guidance for long-term prescription is imperative.

High intensity interval training (HIIT) describes exercise that is characterised by short bursts of vigorous effort followed by periods of rest or low intensity exercise. High intensity interval trainingis an extremely variable mode of exercise with sessions altered by intensity, duration and number of intervals as well as the duration and activity chosen during the rest period. High intensity interval training has been shown to be an effective alternative to traditional endurance training so often used in exercise interventions. It has also been suggested that High intensity interval trainingis more enjoyable than moderate intensity exercise. These findings are important because lack of time and lack of enjoyment are two of the most commonly quoted barriers to regular activity.

The project utilises a pre-experimental one-group pre-test - post-test design. The participants will be assessed at baseline, followed by an intervention and then measured again at follow up.Patients will be purposively recruited from the multiple sclerosis clinic at the Royal Hallamshire Hospital in Sheffield. Potential participants will be identified by consultant neurologists to the research assistant from clinic lists/patient records. Patients who satisfy the inclusion and exclusion criteria will be given/sent a recruitment letter and participant information sheet informing them about the study. The letter will contain a tear-off slip for patients to return to the research team indicating their interest or not in study participation. It will be clearly stated in the letter that there is no obligation or pressure to participate and that if patients are not interested their future medical care will not be jeopardised. Patients who respond to the letter of invitation will be invited into the Centre for Sport and Exercise Science for a consultation.

Once a participant has been recruited and provided informed consent they will attend a baseline assessment. Each participant will undergo a VO2peak test on a cycle ergometer. Gas measurement will be conducted breath by breath by means of telemetric spirometry, heart rate will be measured by Polar system. The test will be conducted to volitional exhaustion or will be terminated when any of the following criteria are met:

* symptom exacerbation
* symptoms indicating risk for the safety or health of the patients
* plateau in oxygen uptake with increasing workload and/ or
* respiratory exchange rate greater than 1.15

Three questionnaires will be administered to the participants to determine the effects of the exercise interventions on physical activity level (Godin Leisure Time Questionnaire), fatigue (modified fatigue impact scale), and health perception (SF-36). Participants will also be given an ActiGraph accelerometer to wear for 7-days. The procedures will be repeated at follow up by a blinded assessor.

Participants will attend two sessions per week for the 6 week intervention. Each session will consist of 6-10 sets of 60 second high intensity intervals interspersed with 60 seconds recovery. The workload during each interval will be set at 80-90% of peak power achieved during the VO2peak test. This is predicted to elicit 85-95% heart rate reserve in the participants. After each interval the participant's heart rate and rate of perceived exertion (RPE) will be collected. After each session a researcher will complete an Adverse Event form to record if an event occurred or not. Additionally the participant will complete a physical activity enjoyment (Perceived activity enjoyment scale) after one session per week.

Outcomes will be assessed at two-time-points: baseline and after the 6-week intervention. Personal characteristics (e.g. postcode, marital status ethnicity, etc.) and condition specific data (e.g. time since diagnosis, medication, onset of symptoms, use of health care resources etc.) will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of MS more than three months
* EDSS score of less than 2.5
* Aged 18-65
* No more than one relapse in the last 2 years
* Participants on disease modifying therapy (Interferon and Grateramer Acetate) must have been stable on this treatment for at least 3 months prior to entering the study

Exclusion Criteria:

* Failure to meet any of the inclusion criteria
* Experiencing illness or injury that impairs their ability to be physically active
* Living more than 20 miles away from Centre for Sport and Exercise Science

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-04-21 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11-08 (Actual)

PRIMARY OUTCOMES:
Number of participants recruited to the study who adhere to high intensity interval training intervention | 12 months
  Adherence will be measured through attendance to the exercise sessions and compliance to the prescribed intensity
Number of participants with treatment related adverse events as recorded by the research team | 12 months
  The research team will complete an adverse event form after each session, stating whether any adverse events occurred or not. For additional safety monitoring participants will be given a diary to record how they feel immediately after the exercise session, several hours after and the next day.

SECONDARY OUTCOMES:
Physical fitness | baseline and at 6 weeks which is study completion
  changes to physical fitness will be measured using the VO2peak cycle ergometer test
Impact of treatment intervention on multiple sclerosis | baseline and at 6 weeks which is study completion
  Number of Participants with Adverse Events That Are Related to Treatment intervention
Impact of treatment intervention on multiple sclerosis | baseline and at 6 weeks which is study completion
  Number of participants who record changes on the quality of life questions due to the impact of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Basil Sharrack, Professor, Principal Investigator — Sheffield Teaching Hospitals NHS FT
Locations (2):
- United Kingdom (2):
  - Sheffield Hallam University, Sheffield, South Yorkshire
  - Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No